CLINICAL TRIAL: NCT01662700
Title: An Open Label Randomized Comparison of Two Antimalarial Drugs Regimens in Patient With Plasmodium Vivax Malaria in Thailand
Brief Title: Comparison of Two Antimalarial Drugs Regimens in Patient With Plasmodium Vivax Malaria in Thailand
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FTM1202
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Acute Uncomplicated Malaria With P.Vivax Infection
Keywords: P. vivax infection; Artesunate; Chloroquine; Primaquine
MeSH Terms: interventions — Artesunate; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AS2 (Experimental): Artesunate 2 mg/kg/day for 5 days Combine with
  * Primaquine 15 mg is given daily for 14 days.
  * Or primaquine 45 mg is given once a week for 8 weeks in G6PD deficiency patients.
  Interventions: Drug: Artesunate
- Chloroquine (Active Comparator): CH25: Chloroquine 25 mg/kg: 15 mg base/kg on the first days (D0), followed by 5 mg base/kg daily on the second and third day (day1-2) (total 25 mg base/ kg).
  Combine with
  * Primaquine 15 mg is given daily for 14 days.
  * Or primaquine 45 mg is given once a week for 8 weeks in G6PD deficiency patients.
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Artesunate
  Arms: AS2
Drug: Chloroquine
  Arms: Chloroquine

SUMMARY:
In Thailand, the proportion of P.vivax infection has now been increasing and is equal to Plasmodium falciparum since 1998. The incidence of P.vivax has recently been reported as 20 per 1000 population per year. Unlike Plasmodium falciparum, P.vivax infection rarely develops into complicated malaria and death is unusual. However, P.vivax has a dormant stage (the hypnozoite) that persists in the human liver and may cause relapse weeks, months, or even years later. Therefore, P.vivax infection is considered to have greater impact on morbidity than mortality, resulting in significant social and economic burden. Moreover, it is very difficult to control P.vivax transmission, because gametocytes appear almost simultaneously with schizonts.

Radical treatment of the infection, therefore, normally consists of a blood schizontocidal course of chloroquine and a course primaquine for the elimination of the hypnozoites as anti-relapse therapy. In Thailand, chloroquine and primaquine have remained the mainstay chemotherapeutics for the treatment of P.vivax for more than 60 years and resistance has not yet been reported . The relapse rates at day 28 are about 50% without primaquine therapy and about 20% with standard primaquine therapy. Relapse has not been observed among patients receiving high dose primaquine therapy (30 mg daily for 14 days).

Since January 2007, the evidence of reduced susceptibility of Plasmodium falciparum to artemisinins in Western Cambodia at Thai-Cambodia border was first presented and confirmed in a subsequent detailed pharmacokinetic-pharmacodynamic study. Nevertheless, a trend of gradual decline of in vitro sensitivity to chloroquine has been documented in some areas of the country, particularly Thai-Myanmar border. There has been no clinical-parasitological evidence of chloroquine resistant P.vivax in Thai-Cambodia border, Thailand.

The objectives of the present study are to assess in vivo efficacy of first line regimen of chloroquine given with primaquine, and in vitro susceptibility of P.vivax isolates in areas along Thai-Cambodia border, Thailand.

DETAILED DESCRIPTION:
Plasmodium vivax affects 70-80 million cases of malaria worldwide annually, is the major cause of human malaria in parts of Pacific region and South America. In Thailand, the proportion of P.vivax infection has increased and it is now equal to Plasmodium falciparum since 1998. The incidence of P.vivax has recently been reported as 20 per 1000 population per year. Unlike Plasmodium falciparum, P.vivax infection rarely develops into complicated malaria and death is unusual. However, P.vivax has a dormant stage (the hypnozoite) that persists in the human liver and may cause relapse weeks, months, or even years later. Therefore, P.vivax infection is considered to have greater impact on morbidity than mortality, resulting in significant social and economic burden. Moreover, it is very difficult to control P.vivax transmission, because gametocytes appear almost simultaneously with schizonts.

Radical treatment of the infection, therefore, normally consists of a blood schizontocidal course of chloroquine and a course primaquine for the elimination of the hypnozoites as antirelapse therapy. However, chloroquine-resistant P.vivax (CRPv) has been emer-ging in different parts of the world. The first report of chloroquine resistant Plasmodium vivax was in 2 Australian soldiers returning from Papua New Guinea in Indonesia and is now spreading over Asia and the Pacific region. In Thailand, chloroquine and primaquine have remained the mainstay chemotherapeutics for the treatment of P.vivax for more than 60 years and resistance has not yet been reported. Occasional failure of the standard primaquine therapy (15 mg daily for 14 days) to prevent relapse has been observed. However, primaquine resistance has not been confirmed. In Thailand, the relapse rates at day 28 are about 50% without primaquine therapy, and about 20% with standard primaquine therapy. Relapse has not been observed among patients receiving high dose primaquine therapy (30 mg daily for 14 days).

A number of factors are reportedly associated with relapse, or the reappearance of P.vivax, including inadequate primaquine dosage, high parasitaemia at diagnosis, and short duration of symptoms prior to diagnosis, presence of gametocytes on admission, age, and gender. Because the radical cure of P.vivax hypnozoites requires 14 days of primaquine therapy, adherence to the drug regimen may greatly affect the prevention of relapse. Unfortunately, the effect of patient adherence on 14 day primaquine treatment, and its relation to preventing parasite reappearance, is not well-document.

Since January 2007, the evidence of reduced susceptibility of Plasmodium falciparum to artemisinins in Western Cambodia at Thai_Cambodia border was first presented and confirmed in a subsequent detailed pharmacokinetic-pharmacodynamic study. Nevertheless, a trend of gradual decline of in vitro sensitivity to chloroquine has been documented in some areas of the country, particularly Thai-Myanmar border. There has been no clinical-parasitological evidence of chloroquine resistant P.vivax in Thai-Cambodia border, Thailand.

The objectives of the present study are to assess in vivo efficacy of first line regimen of chloroquine given with primaquine, and in vitro susceptibility of P.vivax isolates in areas along Thai-Cambodia border, Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged from 18 years to 65 years old who can come to the study hospital for follow up in case of re-infection
* Acute uncomplicated malaria with P.vivax infection, confirmed by positive blood smear with asexual forms of P. vivax with parasitaemia > 1,000 parasites/microliters
* Fever defined as temperature > 37.5 degree celsius or a history of fever within the last 24 hours
* Written informed consent
* Willingness and ability of the patients/guardians to comply with the study protocol for the duration of the study
* Communicate with Thai language

Exclusion Criteria:

* Mixed infection with other plasmodium species
* For females: pregnancy, breast feeding
* History of allergy or known contraindication to chloroquine, artesunate or primaquine
* Any criteria of severe / complicated malaria (WHO 2010)
* Presence of febrile condition caused by disease other than malaria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Parasite Clearance Rate | 7 days
  Parasite clearance rate as defined by the slope of the linear portion of the natural logarithm parasite clearance curve
Relapse rate of P. vivax | 3 months
  Incidence of relapse in P.vivax infection

SECONDARY OUTCOMES:
Parasite clearance time | 7 days
  Parasite clearance time assessed by microscopy
Parasite density time | 7 days
  Time of parasite count to fall to 50%, 90% and 99% of initial parasite density
Fever clearance time | 7 days
  Fever clearance time (i.e. the time taken for temperature to fall below 37 degrees celsius and remain there for at least 24 hrs)
Proportion of patients with gametocytemia | 7 days
  Proportion of patients with gametocytemia before, during and after treatment, assessed at admission, on day 3 stratified by presence of gametocytes at enrolment
In vitro antimalarial drug susceptibility | 7 days
  IC0, IC90, IC99 of Plasmodium vivax responses to antimalarial drugs ( ex vivo)

CONTACTS AND LOCATIONS:
Locations (4):
- Thailand (4):
  - Khunhan Hospital, Si Sa Ket, Changwat Si Sa Ket
  - Kraburi Hospital, Ranong
  - Phusing Hospital, Si Sa Ket
  - Kap Choeng Hospital, Surin